CLINICAL TRIAL: NCT02505074
Title: Natural History of Melody Valve in the Mitral and Tricuspid Position
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); Children's Hospital and Medical Center (Unknown); University of California, San Francisco (Other); NewYork Presbyterian Hospital (Unknown); The Monroe Carell Jr. Children's Hospital at Vanderbilt (Unknown); Northwell Health (Other); Primary Children's Hospital (Other); Seattle Children's Hospital (Other); Gruppo Ospedaliero San Donato (Unknown); University Hospital Munich (Other); University Children's Hospital, Zurich (Other); Fondation IUCPQ (Other); Hospital for Sick Kids (Unknown)
Responsible Party: Principal Investigator, Sitaram Emani, Cardiovascular Surgeon, Boston Children's Hospital
Other Study IDs: IRB-P00015805
Record Dates: First submitted 2015-06-29; First posted 2015-07-22 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Diseases of Mitral Valve; Tricuspid Valve Disorder
Keywords: mitral valve; tricuspid valve; Melody valve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mitral Valve Replacement: Review of retrospective data of those patients who have had surgical replacement of the mitral valve with the Melody valve.
  Interventions: Procedure: Valve replacement with the Melody valve
- Tricuspid Valve Replacement: Review of retrospective data of those patients who have had surgical replacement of the tricuspid valve with the Melody valve.
  Interventions: Procedure: Valve replacement with the Melody valve

INTERVENTIONS:
Procedure: Valve replacement with the Melody valve — This study will only review patients who have had the Melody valve surgically inserted into the Mitral and/or Tricuspid positions. We will not be reviewing any other intervention type.

SUMMARY:
The Melody valve has historically been used for pulmonary valve replacements; however it has been more recently used in the mitral and tricuspid positions. This multi-center, retrospective, observational study will review the durability of the Melody valve inserted into the mitral or tricuspid positions.

Patients who have undergone Melody valve insertion into either the mitral or tricuspid positions prior to December, 2014 will be eligible for the study. Basic de-identified patient demographics will be collected as well as select clinical data. Ventricular function and valvar function of the affected valve will be retrospectively reviewed both prior to surgery and following, as well as review of operative data. The investigators will also review the most recent follow up data and any subsequent re-interventions on the Melody valve. Data from all sites will be entered into an external REDCap database, using only de-identified data.

DETAILED DESCRIPTION:
Prior to recent advancement in using the Melody valve for atrioventricular valve replacement, there have only been fixed diameter valve options for severe valve disease requiring replacement. This presents numerous obstacles for those pediatric patients who require replacement early in life, as the fixed diameter does not offer options for expansion for somatic growth, and early reoperation will be required.

The Melody valve has been approved for transcatheter implantation into the RVOT (right ventricular outflow tract), and has shown competence within a range of sizes. Recent studies conducted at Boston Children's Hospital of off-label use of the Melody valve into atrioventricular valve positions have shown acceptable short-term valve performance, and that subsequent catheter-based expansion is feasible.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have had a Melody valve inserted into either mitral or tricuspid positions via surgical intervention

Exclusion Criteria:

* There are no exclusion criteria.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who have had a Melody valve inserted via surgical intervention prior to December, 2014, into either the mitral or tricuspid positions, will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Long term durability of Melody Valve in mitral and tricuspid positions, to be measured by degree of stenosis in Melody valve | up to 5 years
Long term durability of Melody Valve in mitral and tricuspid positions, to be measured by grade of regurgitation in Melody valve | up to 5 years
Long term durability of Melody Valve in mitral and tricuspid positions, to be measured by number of necessary re-interventions of Melody valve | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sitaram Emani, MD, Principal Investigator — Cardiovascular Surgeon

REFERENCES:
- [Background] Quinonez LG, Breitbart R, Tworetsky W, Lock JE, Marshall AC, Emani SM. Stented bovine jugular vein graft (Melody valve) for surgical mitral valve replacement in infants and children. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1443-9. doi: 10.1016/j.jtcvs.2013.10.059. Epub 2013 Dec 10. PMID 24332108
- [Background] Hasan BS, McElhinney DB, Brown DW, Cheatham JP, Vincent JA, Hellenbrand WE, Jones TK, Zahn EM, Lock JE. Short-term performance of the transcatheter Melody valve in high-pressure hemodynamic environments in the pulmonary and systemic circulations. Circ Cardiovasc Interv. 2011 Dec 1;4(6):615-20. doi: 10.1161/CIRCINTERVENTIONS.111.963389. Epub 2011 Nov 9. PMID 22075926
- [Background] Kaza AK, Lim HG, Dibardino DJ, Bautista-Hernandez V, Robinson J, Allan C, Laussen P, Fynn-Thompson F, Bacha E, del Nido PJ, Mayer JE Jr, Pigula FA. Long-term results of right ventricular outflow tract reconstruction in neonatal cardiac surgery: options and outcomes. J Thorac Cardiovasc Surg. 2009 Oct;138(4):911-6. doi: 10.1016/j.jtcvs.2008.10.058. Epub 2009 Jul 26. PMID 19660342
- [Derived] Pluchinotta FR, Piekarski BL, Milani V, Kretschmar O, Burch PT, Hakami L, Meyer DB, Jacques F, Ghez O, Trezzi M, Carotti A, Qureshi SA, Michel-Behnke I, Hammel JM, Chai P, McMullan D, Mettler B, Ferrer Q, Carminati M, Emani SM. Surgical Atrioventricular Valve Replacement With Melody Valve in Infants and Children. Circ Cardiovasc Interv. 2018 Nov;11(11):e007145. doi: 10.1161/CIRCINTERVENTIONS.118.007145. PMID 30571200